CLINICAL TRIAL: NCT03408977
Title: Factors That Determine the Responses to Meal Ingestion: Sex Differences
Brief Title: Meal Enjoyment and Tolerance: Sex Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PR(AG)338/2016E
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: meal ingestion; meal tolerance; postprandial responses; hedonic sensations; homeostatic sensations

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men (Experimental)
  Interventions: Other: probe meal
- Women (Experimental)
  Interventions: Other: probe meal

INTERVENTIONS:
Other: probe meal — The probe meal will be served in 150 Kcal portions (10 g foie, 10 g cheese, 5 g chips, 2 g peanuts, 3 g toast, and 27 mL soft drink) up to the level of maximal satiation.

SUMMARY:
Aim: to determine the effect of gender on the responses to meal ingestion. Participants (10 men and 10 women) will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the test meal will be administered 4 h after breakfast. Studies will be conducted in a quiet, isolated room with participants sitting on a chair. Participants will ingest a probe meal up to the level of maximal satiation. The probe meal will be served stepwise (150 Kcal every 5 min). Perception of homeostatic (hunger/satiation, fullness) and hedonic (digestive well-being, mood) sensations will be measured at 5 min intervals 10 min before, during and 20 min after ingestion at 10 min intervals.

ELIGIBILITY:
Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2018-01-08 (Actual)

PRIMARY OUTCOMES:
Meal tolerance | 100 min
  Amount of meal (Kcal) consumed up to the level of maximal satiation (score 5 on a - 5 to + 5 score hunger/satiation scale).

SECONDARY OUTCOMES:
Change in digestive well-being induced by the probe meal | 1 day
  Change in well-being measured by 10 score scales during and after the probe meal.
Change in fullness sensation induced by the probe meal | 1 day
  Change in fullness sensation measured by 10 score scales during and after the probe meal.
Change in mood induced by the probe meal | 1 day
  Change in mood measured by 10 score scales during and after the probe meal.
Change in abdominal discomfort induced by the probe meal | 1 day
  Change in abdominal discomfort measured by 10 score scales during and after the probe meal.
Change in hunger/satiety induced by the probe meal | 1 day
  Change in hunger/satiety measured by 10 score scales during and after the probe meal.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain